CLINICAL TRIAL: NCT02036723
Title: Multicentre Double Blind Randomized Clinical Study Evaluating The Efficacy and Safety of BCD-021 (CJSC BIOCAD, Russia) and Lucentis® (Novartis Pharmaceuticals Canada Inc.) in Patients With Neovascular Wet Age-related Macular Degeneration
Brief Title: Safety and Efficacy Study of BCD-021 Compared to Lucentis® in Patients With Neovascular Wet Age-related Macular Degeneration
Acronym: GALATIR
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GALATIR/BCD-021-3; GALATIR
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Macular Degeneration; Eye Diseases; Neovascular Macular Degeneration; Choroidal Neovascularization; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Choroidal Neovascularization; Geographic Atrophy | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BCD-021 (Experimental): BCD-021 is a product code for bevacizumab biosimilar manufactured by CJSC BIOCAD, Russia.
  In this arm 72 patients will receive BCD-021 at a dose 1.25 mg (in 0.05 ml of solution) as an intravitreal injection on day 1 and then every 28 days during 12 months.
  Interventions: Drug: Bevacizumab
- Lucentis® (Active Comparator): Lucentis® is ranibizumab drug produced by Novartis Pharmaceuticals Canada Inc. In this arm 36 patients will receive Lucentis® at a dose 0.50 mg (in 0.05 ml of solution) as an intravitreal injection on day 1 and then every 28 days during 12 months.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive bevacizumab at a dose 1.25 mg (in 0.05 ml of solution) as an intravitreal injection on day 1 and then every 28 days during 12 months.
  Other Names: BCD-021
  Arms: BCD-021
Drug: Ranibizumab — Patients will receive ranibizumab at a dose 0.50 mg (in 0.05 ml of solution) as an intravitreal injection on day 1 and then every 28 days during 12 months.
  Other Names: Lucentis®
  Arms: Lucentis®

SUMMARY:
GALATIR is a double blind randomized clinical trial comparing efficacy and safety of BCD-021 (bevacizumab) and Lucentis® (ranibizumab) in patients with neovascular wet age-related macular degeneration. The purpose of the study is to demonstrate the non-inferiority of efficacy and safety of BCD-021 compared to Lucentis®.

ELIGIBILITY:
Inclusion Criteria:

* Having signed a written informed consent form;
* Men and women;
* Patients must be from 50;
* Wet AMD in the study eye, defined as: Not previously treated active choroidal neovascular membrane (CNV), including retinal angiomatous proliferation (RAP), with oedema involving the fovea as demonstrated with optical coherence tomography (OCT) and fluorescein angiography (FA). FA shall not be older than 14 days at randomization;
* Best corrected VA for the studied eye ranging between 20/32 (6.3/10) and 20/320 (0.6/10) with EDTRS scale;
* Size of lesion < 12 disk area;
* In case of occult neovessels, proof required of recent development of the lesion: loss of VA of at least 5 letters EDTRS (equivalent one line) in the last 3 months OR appearance of a subretinal hemorrhage OR increase in the size of the lesion (> 10%) using fluorescein angiography during the last month by comparison with the last 3 months OR appearance of OCT criteria of macular oedema type, serous separation of neuro-epithelium, separation of the pigmented epithelial during the last month;
* Only one eye of each study patient may be recruited into the study. If the non-study eye is being treated with anti-VEGF therapy, or develops wet AMD, then the same drug being used in the study eye shall be used in the non-study eye. Treatment must be given double-blind in the non-study eye as well;
* Patient's ability (in Investigator's opinion) to follow the protocol procedures;
* Male and female patients with normal reproductive function and their sexual partners are aware and willing to use voluntarily reliable methods of contraception during the whole period of the study including the screening period. This requirement does not apply to patients who underwent operative sterilization or those defined as post-menopausal (confirmed by medical history documentation) within last 2 years. Reliable methods of contraception suggest using 1 barrier method in combination with 1 of the following methods: spermicides, intra-uterine device etc.

Exclusion Criteria:

* Previous or current treatment with intravitreal injection of an anti-VEGF drug (ranibizumab, bevacizumab, aflibercept or pegaptanib, etc.) in the studied eye;
* Other healing treatment in the studied eye during the last 3 months before the first injection;
* Former vitrectomy in the study eye;;
* Medical history of photocoagulation in the studied eye;
* Involvement in another clinical study (studied eye and/or the other eye);
* Subretinal haemorrhage reaching the fovea centre, with a size > 50% of the lesion area;
* Fibrosis or retrofoveal retinal atrophy in the studied eye;
* Retinal pigment epithelial tear reaching the macula in the studied eye;
* Choroidal neovascularisation not related to a AMD in the studied eye;
* Medical history of intravitreal medical device in the studied eye;
* Active or suspected ocular or peri-ocular infection;
* Acute conjunctivitis, keratitis, scleritis, or endophthalmitis;
* Serious active intra-ocular inflammation in the studied eye;
* Macula-foramen of the studied eye;
* Myopia larger than -8 diopter;
* Former corneal grafting of the studied eye;
* Medical history of auto-immune or idiopathic uveitis;
* Proved diabetic retinopathy;
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments;
* Medical history of intra-ocular surgery within 2 months before the first injection in the studied eye;
* Aphakia or lack of lens capsule (not removed by laser) in the studied eye;
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion;
* Known hypersensitivity to ranibizumab, bevacizumab, or another drug composite of the medicinal products used; allergy to fluorescein, indocyanine green, anaesthetic eye drops;
* Arterial hypertension that is not controlled by an appropriate treatment;
* Previous or current treatment with systemic administration of bevacizumab;
* Pregnancy and breast-feeding;
* Any determined immunodeficiency;
* Syphilis, HIV, hepatitis B, any history of hepatitis C virus;
* Any mental disorder, including major depression and/or suicidal thoughts in anamnesis that can, in Investigator's opinion, create a risk for the patient or influence the patient's ability to follow the study protocol;
* Drug addiction, alcoholism.
* Presence or history of malignant neoplasm (including lymphoproliferative disease), with the exception of: Adequately treated basal cell carcinoma and cervical carcinoma in situ; Any malignancy with complete remission of more than 5 years;
* Simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation; previous participation in this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
• Proportion of patients losing fewer than 15 letters on EDTRS chart at month 12 | week 52

SECONDARY OUTCOMES:
• Frequency of ocular and systemic adverse events (AE) and serious adverse events (SAE) that are related, in Investigator's opinion, to AMD therapy | week 52
• Frequency of AE and SAE with toxicity level of 3-4 that are related, in Investigator's opinion, to AMD therapy | week 52
• Number of cases of early withdrawal from the study caused by AE or SAE | week 52
• Number of patients who have binding and neutralizing antibodies to BCD-021/Lucentis in serum at screening and month 12 | screening, week 52
• The mean titer of binding and neutralizing antibodies to BCD-021/Lucentis in serum at screening and month 12 | screening, week 52
• Mean change in VA score, measured on the EDTRS scale at month 12 | week 52
• Average number of injections and time before re-injection | week 52
• Lesion size at month 6 and month 12 (by angiography) | week 26, 52
• Lesion leakage at month 6 and month 12 | week 26, 52
• Change in fluid and foveal thickness on OCT during the study | week 52
• Retinal sensitivity measured by microperimetry at screening, at month 6 and month 12 | screening, week 26, 52
• Timing of visual improvement after initiation of therapy | week 52

CONTACTS AND LOCATIONS:
Locations (13):
- Brazil (7):
  - Hospital dos Olhos do Paraná, Curitiba, Paraná
  - Universidade Estadual de Londrina, Londrina, Paraná
  - Universidade Federal de Minas Gerais Hospital das Clínicas, Belo Horizonte
  - UERJ Hospital Universitário Pedro Ernesto, Rio de Janeiro
  - Universidade Federal do Rio de Janeiro Hospital Clementino Fraga Filho, Rio de Janeiro
  - Universidade de São Paulo Faculdade de Medicina de Ribeirão Preto, São Paulo
  - Universidade Federal de São Paulo Hospital São Paulo, São Paulo
- Russia (6):
  - Republican Clinical Eye Hospital, Kazan', Tatarstan Republic
  - Scientific and Research Institute named after Helmholtz, Moscow
  - IRTC "Eye Microsurgery" named after academician SN Fedorov ", Saint Petersburg
  - Municipal Advisory and Diagnostic Centre number 1, Saint Petersburg
  - St. Petersburg State Medical University named after academician IP Pavlova, Saint Petersburg
  - Regional Clinical Ophthalmic Hospital named TI Yeroshevsky, Samara